CLINICAL TRIAL: NCT01048658
Title: Sevoflurane as an Anesthetic During Dilation and Evacuation Procedures: Does it Increase Blood Loss and Interventions for Blood Loss and Why Do Anesthesiologists Choose to Use It?
Brief Title: Sevoflurane as an Anesthetic During Dilation and Evacuation Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Rosanne Botha, Master of Public Health Student, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB - 5146
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Blood Loss; Anesthesia
Keywords: Sevoflurane; anesthesia; abortion; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Active Comparator): Subject receives Sevoflurane in addition to other standard of care drug regimens for anesthesia with this procedure.
  Interventions: Drug: Sevoflurane
- No Sevoflurane (Placebo Comparator): Subject receives standard of care drug regimens for anesthesia with this procedure.
  Interventions: Other: No Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Subject receives Sevoflurane in addition to other standard of care drug regimens for anesthesia with this procedure.
  Other Names: Ultane
  Arms: Sevoflurane
Other: No Sevoflurane — Subject only standard of care drug regimens for anesthesia with this procedure.
  Arms: No Sevoflurane

SUMMARY:
Sevoflurane is an FDA-approved anesthetic drug commonly used for anesthesia during second trimester abortion procedures. It has a few advantages, including ease of use by the anesthesia provider. However, the literature suggests that when used in doses higher than those used at Oregon Health & Science University (OHSU) and Lovejoy, it is associated with an increase in the risk of bleeding. The investigators study aims to test whether the lower dose used at OHSU and Lovejoy during second trimester abortion procedures causes any difference in blood loss, when compared to similar abortion procedures for which this drug is not used.

DETAILED DESCRIPTION:
This study seeks to examine the bleeding complications associated with use of sevoflurane in general anesthesia regimens for second trimester abortion procedures and assess anesthesia providers' use and beliefs regarding possible risks associated with newer inhalational agents such as sevoflurane in this setting. Participants' anesthesia will either be intravenous (IV) propofol, IV midazolam, IV fentanyl and nitrous oxide or this same regimen combined with sevoflurane during maintenance of anesthesia. Procedural outcomes, specifically those related to bleeding complications, including need to intervene for excess blood loss, will be recorded and analyzed to establish if such a relationship between use of sevoflurane and excess blood loss exists.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily requesting pregnancy termination
* Estimated gestational age of 18 weeks - 23 weeks, 6 days gestational age as calculated by fetal biparietal diameter on clinic ultrasound.
* Be able and willing to sign an informed consent and agree to terms of the study

Exclusion Criteria:

* Known severe maternal respiratory disease or upper respiratory infection or sinus blockage
* Anticoagulation use: within 24 hours if Lovenox, or within 12 hours if heparin, (Must have a documented normal international normalized ratio (INR) prior to procedure if on anticoagulation)
* Multiple pregnancy
* Fetal demise, if more than 2 weeks difference exists between known gestational age (by previous US dating) and gestational size on current ultrasound.
* Known allergy/sensitivity to sevoflurane or any other inhaled anesthetic agents

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosanne Botha, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Lovejoy Surgicenter, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon

REFERENCES:
- [Background] Socio-Economic Factbook, S.A. Department, Editor. 1993, American College of Surgeons: Chicago, IL.
- [Background] Paul, M., A Clinician's Guide to Medical and Surgical Abortion. 1999, New York, New York: Church Livingstone.
- [Background] Peterson WF, Berry FN, Grace MR, Gulbranson CL. Second-trimester abortion by dilatation and evacuation: an analysis of 11,747 cases. Obstet Gynecol. 1983 Aug;62(2):185-90. PMID 6866362
- [Background] Method, weeks of gestation key in abortion complications. Contracept Technol Update. 1980 Oct;1(7):96-7. PMID 12336808
- [Background] MacKay HT, Schulz KF, Grimes DA. Safety of local versus general anesthesia for second-trimester dilatation and evacuation abortion. Obstet Gynecol. 1985 Nov;66(5):661-5. PMID 4058825
- [Background] O'Connell K, Jones HE, Lichtenberg ES, Paul M. Second-trimester surgical abortion practices: a survey of National Abortion Federation members. Contraception. 2008 Dec;78(6):492-9. doi: 10.1016/j.contraception.2008.07.011. Epub 2008 Sep 4. PMID 19014796
- [Background] Abboud TK, D'Onofrio L, Reyes A, Mosaad P, Zhu J, Mantilla M, Gangolly J, Crowell D, Cheung M, Afrasiabi A, et al. Isoflurane or halothane for cesarean section: comparative maternal and neonatal effects. Acta Anaesthesiol Scand. 1989 Oct;33(7):578-81. doi: 10.1111/j.1399-6576.1989.tb02970.x. PMID 2816239
- [Background] West SL, Moore CA, Gillard M, Browne PD. Anaesthesia for suction termination of pregnancy. Anaesthesia. 1985 Jul;40(7):669-72. doi: 10.1111/j.1365-2044.1985.tb10948.x. PMID 4025771
- [Background] Collins KM, Plantevin OM, Whitburn RH, Doyle JP. Outpatient termination of pregnancy: halothane or alfentanil-supplemented anaesthesia. Br J Anaesth. 1985 Dec;57(12):1226-31. doi: 10.1093/bja/57.12.1226. PMID 3936528
- [Background] Forrest WH Jr. Effects of anesthesia in therapeutic abortion. Anesthesiology. 1970 Jul;33(1):121-2. doi: 10.1097/00000542-197007000-00028. No abstract available. PMID 4393415
- [Background] Cullen BF, Margolis AJ, Eger EI 2nd. The effects of anesthesia and pulmonary ventilation on blood loss during elective therapeutic abortion. Anesthesiology. 1970 Feb;32(2):108-13. doi: 10.1097/00000542-197002000-00004. No abstract available. PMID 4391841
- [Background] Patel SS, Goa KL. Sevoflurane. A review of its pharmacodynamic and pharmacokinetic properties and its clinical use in general anaesthesia. Drugs. 1996 Apr;51(4):658-700. doi: 10.2165/00003495-199651040-00009. PMID 8706599
- [Background] Yamakage M, Tsujiguchi N, Chen X, Kamada Y, Namiki A. Sevoflurane inhibits contraction of uterine smooth muscle from pregnant rats similarly to halothane and isoflurane. Can J Anaesth. 2002 Jan;49(1):62-6. doi: 10.1007/BF03020420. PMID 11782330
- [Background] Turner RJ, Lambrost M, Holmes C, Katz SG, Downs CS, Collins DW, Gatt SP. The effects of sevoflurane on isolated gravid human myometrium. Anaesth Intensive Care. 2002 Oct;30(5):591-6. doi: 10.1177/0310057X0203000508. PMID 12413258
- [Background] Nathan N, Peyclit A, Lahrimi A, Feiss P. Comparison of sevoflurane and propofol for ambulatory anaesthesia in gynaecological surgery. Can J Anaesth. 1998 Dec;45(12):1148-50. doi: 10.1007/BF03012454. PMID 10051930
- [Background] Nelskyla K, Korttila K, Yli-Hankala A. Comparison of sevoflurane-nitrous oxide and propofol-alfentanil-nitrous oxide anaesthesia for minor gynaecological surgery. Br J Anaesth. 1999 Oct;83(4):576-9. doi: 10.1093/bja/83.4.576. PMID 10673872
- [Background] Karaman S, Akercan F, Aldemir O, Terek MC, Yalaz M, Firat V. The maternal and neonatal effects of the volatile anaesthetic agents desflurane and sevoflurane in caesarean section: a prospective, randomized clinical study. J Int Med Res. 2006 Mar-Apr;34(2):183-92. doi: 10.1177/147323000603400208. PMID 16749414
- [Background] Gambling DR, Sharma SK, White PF, Van Beveren T, Bala AS, Gouldson R. Use of sevoflurane during elective cesarean birth: a comparison with isoflurane and spinal anesthesia. Anesth Analg. 1995 Jul;81(1):90-5. doi: 10.1097/00000539-199507000-00018. PMID 7598289
- [Background] Toscano A, Pancaro C, Giovannoni S, Minelli G, Baldi C, Guerrieri G, Crowhurst JA, Peduto VA. Sevoflurane analgesia in obstetrics: a pilot study. Int J Obstet Anesth. 2003 Apr;12(2):79-82. doi: 10.1016/S0959-289X(02)00195-4. PMID 15321492
- [Background] Jackson RA, Teplin VL, Drey EA, Thomas LJ, Darney PD. Digoxin to facilitate late second-trimester abortion: a randomized, masked, placebo-controlled trial. Obstet Gynecol. 2001 Mar;97(3):471-6. doi: 10.1016/s0029-7844(00)01148-0. PMID 11239659
- [Background] Turok DK, Gurtcheff SE, Esplin MS, Shah M, Simonsen SE, Trauscht-Van Horn J, Silver RM. Second trimester termination of pregnancy: a review by site and procedure type. Contraception. 2008 Mar;77(3):155-61. doi: 10.1016/j.contraception.2007.11.004. Epub 2008 Jan 11. PMID 18279684

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sevoflurane | No Sevoflurane
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | No Sevoflurane | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (6.2) | 25.9 (5.9) | 25.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Needing Intervention to Treat Blood Loss (a Composite of Use of Uterotonics, Re-aspiration, and Bimanual Massage)
Description: Provider report for need to intervene due to blood loss (yes/no)
Time Frame: At time of uterine evacuation and immediately post-operatively, an average of 7.1 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Sevoflurane | No Sevoflurane
Number analyzed (Participants) | 80 | 80
Participants | 20 | 13

2. Secondary Outcome: Number of Participants With Estimated Blood Loss Greater Than 300 mL (Yes/no)
Description: Procedural blood loss greater than 300 mL. Blood loss was measured in a standardized fashion (amniotic fluid was discarded, blood was separated from tissue, and all gauze surgical drapes weighed).
Time Frame: At time of uterine evacuation, an average of 7.1 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Sevoflurane | No Sevoflurane
Number analyzed (Participants) | 80 | 80
Participants | 12 | 6

3. Secondary Outcome: Procedure Time: T-test (Time of Speculum Placement to Time Speculum Removed)
Description: Length of procedure from time of speculum placement to time of speculum removal, in minutes.
Time Frame: Time of speculum place to time of speculum removal, an average of 7.1 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sevoflurane | No Sevoflurane
Number analyzed (Participants) | 80 | 80
minutes | 7.0 (3.7) | 7.3 (3.3)

4. Secondary Outcome: Number of Participants Experiencing Side Effects (Nausea, Dizziness)
Time Frame: Post-procedure, within 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Sevoflurane | No Sevoflurane
Number analyzed (Participants) | 80 | 80
Participants | 13 | 11

5. Secondary Outcome: Patient and Provider Satisfaction With Anesthesia
Description: Scores reported on 10-cm Visual Analog Scale (VAS anchors: 0= not satisfied at all, 10= completely satisfied) . Reported as mean +/- standard deviation. Subjects and providers were blinded to anesthesia method. Subjects and providers completed post-operative questionnaire within 30 minutes of procedure completion.
Time Frame: Post-procedure, within 30 minutes
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sevoflurane | No Sevoflurane
Number analyzed (Participants) | 80 | 80
cm
  Provider Satisfaction | 9.4 (1.1) | 9.3 (1.4)
  Patient Satisfaction | 8.4 (1.5) | 8.2 (1.5)

ADVERSE EVENTS:
Time Frame: During and post-procedure
Arm/Group | Sevoflurane | No Sevoflurane
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/80
Other Adverse Events (participants affected / at risk) | 3/80 | 1/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevoflurane (N=80) | No Sevoflurane (N=80)
Blood loss and unterine atony (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevoflurane (N=80) | No Sevoflurane (N=80)
Cervical laceration (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Unterine atony (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes